CLINICAL TRIAL: NCT03653663
Title: Near Infrared Spectroscopy to Diagnose Statin-Associated Muscle Symptoms
Brief Title: NIRS to Diagnose SAMS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hartford Hospital (Other)
Collaborators: University of Connecticut (Other)
Responsible Party: Principal Investigator, Beth Taylor, Director of Exercise Physiology Research, Hartford Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: Grant-In-Aid #17GRNT33661247
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Statin Adverse Reaction; Skeletal Myopathy
MeSH Terms: interventions — Simvastatin

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized crossover study of placebo vs. 20 mg simvastatin for 8 weeks with a 4 week washout in between
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All members of the investigative team as well as the patients are blinded to treatment until all subjects have completed the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 8 weeks treatment with placebo (or until muscle symptoms appear for at least 1 week or are unbearable)
  Interventions: Drug: Placebo Oral Tablet
- 20 mg simvastatin (Active Comparator): 8 weeks treatment with 20 mg simvastatin daily (or until muscle symptoms appear for at least 1 week or are unbearable)
  Interventions: Drug: Simvastatin 20 mg

INTERVENTIONS:
Drug: Simvastatin 20 mg — Subjects are treated with 20 mg simvastatin for 8 weeks
  Arms: 20 mg simvastatin
Drug: Placebo Oral Tablet — Subjects are treated with placebo for 8 weeks
  Arms: Placebo

SUMMARY:
This proposal seeks to determine whether near infrared spectroscopy (NIRS) can differentiate between patients with confirmed SAMS and those with non-specific muscle complaints. NIRS is a non-invasive technique of assessing skeletal muscle tissue oxygenation and mitochondrial function. Mitochondrial dysfunction is a possible cause of SAMS, but NIRS has never been evaluated as a diagnostic tool for SAMS. Investigators will enroll 40 patients with a history of SAMS in an 8 wk randomized, double-blind crossover trial of simvastatin 20 mg/d and placebo separated by a 4 wk washout phase. Tissue oxygenation will be measured using NIRS during a short handgrip exercise protocol before and after each treatment period. Investigators will query patients about muscle complaints weekly during both phases of the study with a validated survey to assess muscle pain. Investigators will classify patients as testing positive for SAMS if they report pain on simvastatin and not placebo. Investigators hypothesize that these patients, vs. patients experiencing pain on both treatments, placebo, or neither treatment, will be distinguished by reduced tissue oxygenation during simvastatin treatment relative to placebo, demonstrating efficacy of NIRS as a clinical tool that can be eventually used for the diagnosis and ultimately treatment of SAMS.

DETAILED DESCRIPTION:
Study Overview: Forty patients with possible SAMS will be recruited from the Cholesterol Management Center at Hartford Hospital, advertisements and contact with physicians' offices. Subjects will be withdrawn from all statin lipid lowering medications for at least 4 weeks. Subjects will then undergo baseline testing (tissue oxygenation will be measured using NIRS during a short handgrip exercise protocol) and be randomized to treatment with simvastatin 20 mg daily or matching placebo for up to 2 months. Subjects will be called weekly to assess symptoms of muscle pain and administer the Brief Pain Inventory (BPI). NIRS measurements will be repeated and treatment (simvastatin or placebo) will be stopped after 2 months or after subjects have experienced muscle symptoms continuously for one week. After 4 weeks washout, subjects will again be randomized to simvastatin or placebo treatment and the monitoring and measurement processes will be repeated (see study schematic below). Those patients developing muscle symptoms during statin treatment but not during placebo treatment will be considered to have confirmed SAMS. Investigators hypothesize that patients with confirmed SAMS will be distinguished from all other patients with reduced tissue oxygenation during simvastatin treatment relative to placebo, demonstrating efficacy of NIRS as a clinical tool that can be eventually used for the diagnosis and ultimately treatment of SAMS.

Study Subjects: Statin myopathic symptoms have been poorly defined in the medical literature. For the purpose of this study, investigators will use similar criteria as the previous CoQ10 in Statin Myopathy Study when recruiting eligible subjects. Subjects will be considered to have had prior statin related complaints and recruited for participation in the study if the following occurred: 1) They developed new myalgia, cramps, or muscle aching during statin treatment; 2) The symptoms resolved within 4 weeks of stopping the statin; 3) The identical symptoms recurred during repeat statin exposure. Investigators will recruit men and women ≥40 yrs of age, since older age is a risk factor for SAMS and 25% of U.S. adults ≥40 yrs report statin use. Investigators will enroll equal numbers of men and women to improve the generalizability of the results. Investigators will not exclude individuals with diagnosed coronary artery disease, peripheral vascular disease, or an elevated CK off treatment<10 upper normal limit (UNL) because spontaneous elevations in CK levels are normal in the general population. During the study, subjects will be contacted by phone weekly to inquire about muscle complaints using the Brief Pain Inventory (Short Form) (BPI-SF). Results will be recorded on paper forms and entered into the database. After 1 week of persistent symptoms or as soon as possible if the patient has intolerable symptoms, the subject will undergo NIRS testing and be taken off study drug. This reduces undue subject burden such that subjects do not have to maintain statin treatment for multiple weeks with pain symptoms. Subjects who do not report recurrent symptoms will be treated for 8 weeks, at which time they will undergo 4 weeks washout and move on to the crossover phase. Subjects will be reimbursed $200 for study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects >40 years of age, equal numbers of age, with a prior history of statin-associated muscle symptoms (SAMS). Subjects will be considered to have had prior statin related complaints and recruited for participation in the study if the following occurred: 1) They developed new pain, cramps, or muscle aching during statin treatment; 2) The symptoms resolved within 4 weeks of stopping the statin; 3) The identical symptoms recurred during repeat statin exposure.

Exclusion Criteria:

Subjects who have had cancer within 5 years of entry, have hepatic disease (ALT > 2 times normal) or renal disease (creatinine > 2 mg/L) since these patients may require more careful monitoring during the study and would be best managed in a totally clinical setting

* Subjects presently treated with other medications known to alter statin metabolism;
* Subjects with hypo- or hyperthyroidism defined as a TSH > 5 or <0.01 IU/L since these conditions are known to be associated with statin intolerance and muscle weakness, respectively;1,2
* Subjects with hepatic dysfunction evidenced by a baseline alanine aminotransferase (ALT) level > 2 UNL;1,2
* Subjects with renal dysfunction defined as a baseline creatinine > 2mg/dl;
* Subjects with physical disabilities prohibiting the handgrip protocol;
* Women who are pregnant as determined by a urine pregnancy test using an Accutest Early Pregnancy Test Kit, or who are trying to become pregnant, and/or who have not been using a form of birth control for at least the last 3 months, since the impact of statins on pregnancy-related outcomes has not been well studied;1
* Subjects who regularly use corticosteroids or other drugs known to affect skeletal muscle metabolism or regularly have intramuscular injections that will affect CK levels.

Subjects who are unwilling to limit their alcohol intake to an average of two or less drinks daily.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-02-29 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Near infrared spectroscopy | Up to 8 weeks of treatment, or until muscle symptoms have occurred for 1 week or are intolerable
  Changes in muscle oxygenation with near infrared spectroscopy during incremental handgrip exercise with drug treatment

SECONDARY OUTCOMES:
Creatine kinase | Up to 8 weeks of treatment, or until muscle symptoms have occurred for 1 week or are intolerable
  Changes in creatine kinase with drug treatment

CONTACTS AND LOCATIONS:
Overall Officials: Beth Taylor, PhD, Principal Investigator — Hartford Hospital
Locations (2):
- United States (2):
  - Hartford Hospital, Hartford, Connecticut
  - University of Connecticut, Storrs, Connecticut

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mangone LA, Taylor BA, Schmelzer R, Noh SG, White MC, Kwon OS, Thompson PD. Skeletal muscle mitochondrial capacity in patients with statin-associated muscle symptoms (SAMS). Open Heart. 2024 Feb 22;11(1):e002551. doi: 10.1136/openhrt-2023-002551. PMID 38388189